CLINICAL TRIAL: NCT01434511
Title: Efficacy and Safety of B-Domain Deleted Recombinant Porcine Factor VIII (OBI-1) in the Treatment of Patients With Congenital Hemophilia A With Factor VIII Inhibitors
Brief Title: Study of Modified Recombinant Factor VIII (OBI-1) in Subjects With Congenital Hemophilia A
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBI-1-302
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
Keywords: hemophilia A; haemophilia A; blood coagulation disorders; hemorrhagic disorders; coagulation protein disorder; hematologic diseases; congenital hemophilia A
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Hemorrhagic Disorders; Coagulation Protein Disorders; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OBI-1 (Experimental)
  Interventions: Biological: OBI-1

INTERVENTIONS:
Biological: OBI-1 — intravenous infusion, up to every 2-3 hours for the first 24 hours of treatment

SUMMARY:
This study is to test whether the study drug (OBI-1) is safe and effective for the treatment of serious bleeding episodes in people with congenital hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent from participant and/or participant's parent or legal representative.
* Participants with congenital hemophilia A with human factor VIII inhibitor ≤30 BU assessed within 90 days prior to study entry.
* Has previously or is currently demonstrating suboptimal hemostatic response to bypassing agents for treatment of bleeding episodes; suboptimal response is determined by the investigator , but minimally includes no or minimal evidence of response after at least two doses of bypassing agents, either for the current or a historic bleeding episode.
* Has an anti-OBI-1 titer ≤ 10 BU
* Has any serious or life-threatening bleeding episode; or requires a surgical procedure that could lead to a serious bleeding episode if not well controlled.
* Is willing and able to follow all instructions and attend all study visits.
* Has no other significant hemostatic abnormality and:

  * Platelets ≥100,000/mm-cubed
  * Prothrombin time < 15 seconds
  * INR < 1.3
* Participants taking anti-thrombotics (such as clopidogrel, heparin or heparin analogue) may be included provided three half-lives of the agent have elapsed since the last dose of the agent.

Exclusion Criteria:

* Hemodynamically unstable after blood transfusion, fluid resuscitation and pharmacologic or volume replacement pressor therapy. This hemodynamic instability is characterized by symptomatic hypotension resulting in vital organ dysfunction, such as cardiac ischemia, oliguria (urine volume <0.5 mL/kg in the previous six hours), central nervous system hypoperfusion manifested by mental status change such as confusion (unless head injury or intracranial hemorrhage is present), pulmonary compromise, and/or acidosis (manifested by pH and lactate levels).
* Bleeding episode assessed likely to resolve on its own if left untreated.
* Use of hemophilia medication: recombinant factor VIIa within 3 hours prior to OBI-1 administration or activated prothrombin complex concentrate (aPCC) treatment within 6 hours prior to OBI-1 administration
* Prior history of bleeding disorder other than congenital hemophilia A
* Known major sensitivity (anaphylactoid reactions) to porcine or hamster products. Examples include therapeutics of porcine origin (e.g. previously marketed porcine factor VIII, Hyate-C®) and recombinant therapeutics prepared from hamster cells (e.g. Humira®, Advate® and Enbrel®).
* Received any other investigational treatment within 30 days of the first OBI-1 treatment.
* Anticipated need for treatment or device during the study that may interfere with the evaluation of the safety or efficacy of OBI-1, or whose safety or efficacy may be affected by OBI-1.
* Is planning to father a child during the study
* Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the participant's safety or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
* Inability or unwillingness to comply with the study design, protocol requirements, or the follow-up procedures.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2013-07-29 (Actual); Study Completion 2013-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana, United States
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa
- Great Ormond Street Hospital, London, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OBI-1
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated early and only enrolled one participant. Due to concerns that the participant would be at risk of being re-identified, study results are not posted. The decision to terminate this study was not related to any safety and/or efficacy concern of OBI-1 in the indication described within this study (Congenital Hemophilia A).
Arm/Group | OBI-1
Number analyzed (Participants) | 0
Age, Continuous [unit: years] — This study was terminated early and only enrolled one participant. Due to concerns that the participant would be at risk of being re-identified, study results are not posted. The decision to terminate this study was not related to any safety and/or efficacy concern of OBI-1 in the indication described within this study (Congenital Hemophilia A).
Sex: Female, Male — This study was terminated early and only enrolled one participant. Due to concerns that the participant would be at risk of being re-identified, study results are not posted. The decision to terminate this study was not related to any safety and/or efficacy concern of OBI-1 in the indication described within this study (Congenital Hemophilia A).
Region of Enrollment — This study was terminated early and only enrolled one participant. Due to concerns that the participant would be at risk of being re-identified, study results are not posted. The decision to terminate this study was not related to any safety and/or efficacy concern of OBI-1 in the indication described within this study (Congenital Hemophilia A).

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Serious Bleeding Episodes Responsive to OBI-1
Description: This study was terminated early and only enrolled one participant. Due to concerns that the participant would be at risk of being re-identified, the study results are not posted. The decision to terminate this study was not related to any safety and/or efficacy concern of OBI-1 in the indication described within the OBI-1-302 study (Congenital Hemophilia A).
Time Frame: 24 hours after initiation of treatment
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Proportion of Serious Bleeding Episodes Successfully Controlled With OBI-1 Therapy, as Assessed by the Investigator.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Bleeding Episodes Responsive to OBI-1 Therapy at Designated Assessment Time Points After the Initiation of Therapy, as Assessed by the Investigator
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency of Infusions of OBI-1 Required to Successfully Control Qualifying Bleeding Episodes.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

5. Secondary Outcome: Total Dose of OBI-1 Required to Successfully Control Qualifying Bleeding Episodes.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

6. Secondary Outcome: Total Number of Infusions of OBI-1 Required to Successfully Control Qualifying Bleeding Episodes.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

7. Secondary Outcome: Correlation Between Response to OBI-1 Therapy at Specified Time Points and Eventual Control of Serious Bleeding Episodes.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

8. Secondary Outcome: Correlation Between the Pre-infusion Anti-OBI-1 Antibody Titers, the Total Dose of OBI-1, the Outcome at 24 Hours and the Eventual Control of the Bleeding Episode.
Time Frame: Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlation Between the Pre-infusion Anti-OBI-1 Antibody Titers and the Recovery of OBI-1.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

10. Secondary Outcome: Recovery and Elimination Rate Parameters of OBI-1 in Subjects With Inhibitors Treated With OBI-1 Therapy.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

11. Secondary Outcome: Efficacy Assessment of OBI-1 in Participants With Anti-human Factor VIII Titers >30 Bethesda Units (BU)
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

12. Secondary Outcome: Anti-human Factor VIII Antibody Titer.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

13. Secondary Outcome: Anti-OBI-1 Antibody Titer.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

14. Secondary Outcome: Anti-host Cell Protein Baby Hamster Kidney (BHK) Antibody Titer.
Time Frame: Through 90 days ± 7days following final OBI-1 dose
Population: as for baseline characteristics
Arm/Group | OBI-1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | OBI-1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 12 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥30 days prior to submission or communication. Baxter may request an additional delay of ≤30 days(e.g., for intellectual property protection)